CLINICAL TRIAL: NCT05583864
Title: Lumbar Fusion With Porous Titanium Versus Non-Porous Titanium-Coated PEEK Interbody Cages - A Randomized Controlled Trial
Brief Title: Lumbar Fusion With Porous Versus Non-Porous Cages
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kentucky (Other)
Responsible Party: Principal Investigator, Francis Farhadi, Associate Professor, Neurosurgery, University of Kentucky
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 77018
Record Dates: First submitted 2022-10-13; First posted 2022-10-18 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Spinal Fusion; Lumbar Fusion; Arthrodesis; Spondylolisthesis; Pseudarthrosis
Keywords: Spinal Cage; PEEK; Pseudarthrosis; Spondylolisthesis; Titanium; Fusion; Transforaminal; Interbody; Posterolateral; CONDUIT; PROTI 360; TLIF
MeSH Terms: conditions — Ankylosis; Spondylolisthesis; Pseudarthrosis

STUDY DESIGN:
Intervention Model Description: Two types of spinal cages will be evaluated against one another for patient outcomes. It is possible that a single patient may receive both cages, but outcomes will be radiographically assessed individually by cage.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-Blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- CONDUIT Porous Titanium Spinal Cage (Active Comparator): Solid titanium spinal cage, infused with microscopic, porous canals to allow for adhesion and proliferation of bone graft factors contributing to spinal ossification, and ultimately, spinal fusion between vertebrae demonstrating instability.
  Interventions: Device: CONDUIT Porous Titanium Spinal Cage
- PROTI 360 Titanium-Coated PEEK Spinal Cage (Active Comparator): Spinal cage composed primarily of a medical-grade polymer: poly-ether-ether-ketone (PEEK), with a titanium coating that is etched, but lacking porous features. These design features also attempt to stimulate spinal vertebrae fusion through bone-graft ossification and enhance vertebral stability.
  Interventions: Device: PROTI 360 Titanium-Coated PEEK Spinal Cage

INTERVENTIONS:
Device: CONDUIT Porous Titanium Spinal Cage — Already included in arm/group descriptions.
  Other Names: DePuy Synthes CONDUIT™
  Arms: CONDUIT Porous Titanium Spinal Cage
Device: PROTI 360 Titanium-Coated PEEK Spinal Cage — Already included in arm/group descriptions.
  Other Names: DePuy Synthes PROTI 360º™
  Arms: PROTI 360 Titanium-Coated PEEK Spinal Cage

SUMMARY:
The objective of this single site, randomized controlled trial is to assess and compare radiographic and clinical outcomes in patients who are to undergo lumbar interbody fusion procedures (TLIF), supplemented with pedicle screw instrumentation, using one of the following interventions:

1. Porous titanium cages
2. Non-porous titanium-coated poly-ether-ether-ketone (PEEK) cages.

DETAILED DESCRIPTION:
This single-center randomized controlled trial will prospectively evaluate the safety and efficacy of porous titanium cages supplemented with a pedicle screw system as compared to titanium-coated PEEK cages currently used in routine fashion for lumbar interbody fusion procedures.

These cages are FDA approved and the study is designed to compare the outcomes of subjects receiving either implant. This study will capture clinical and radiographic outcomes on patients up to 2 years post-operatively. Both cages will be used in conjunction with milled local autograft bone generated as part of the spinal fusion procedure (no iliac crest autograft will be utilized).

This study will enroll a maximum of 108 subjects (approximately n = 54 per group), with subjects followed for a minimum of 12 months post-surgery. A total cage sample size of 108 cages (n = 54 cages per group) was calculated with a power of 80% (alpha =0.05) and based on the assumption that 55% of cages in the titanium-coated PEEK group would achieve a solid fusion by 6 months, as compared to 80% in the porous titanium group. Up to two cages may be placed in a single subject. Therefore, it is possible that the maximum number of human subjects would be 54 if all are multi-level procedures. Since there are always mixtures of single and multi-level procedures, the actual number of subjects will be closer to 80, with a maximum ceiling of 108.

These assumptions are based on prior imaging findings in patients undergoing TLIF procedures using these cages. An interim analysis is planned once, at minimum, half of the cage accrual is met. In the case early findings show a statistical difference in the primary outcome between the two cages, enrollment will be allowed to cease as investigators are unlikely to maintain clinical equipoise to continue randomizing patients. Conversely, if the interim analysis suggests that statistical significance is unlikely, the investigators will be allowed to choose to close the trial early for futility.

Randomization will occur in 4 and 6 subject blocks to ensure comparability and enhance blinding for this sample size. Subjects will be further stratified for smoking due to the significant risk it places on successful fusion outcomes.

ELIGIBILITY:
Inclusion Criteria:

Patients will be considered for inclusion if:

1. They are scheduled to undergo combined interbody and posterolateral spinal fusion surgery using either the DePuy Synthes CONDUIT™ porous titanium cage or the DePuy Synthes PROTI 360º™ non-porous titanium-coated PEEK cage in conjunction with local autograft bone, and supplementation with a pedicle screw system.
2. They are over the age of 18 years old.
3. They have been unresponsive to conservative care for a minimum of 6 months.
4. They are in the investigator's opinion, be psychosocially, mentally, and physically able to fully comply with this protocol including the required follow-up visits, the filling out of required forms, and have the ability to understand and give written informed consent.

Exclusion Criteria:

Certain comorbidities and medical statuses may render patients ineligible for surgery, or put them at an increased risk for complications or injury by participating in the study. Therefore, patients will be excluded from enrollment if:

1. They have had previous lumbar arthrodesis surgery.
2. They require additional bone grafting materials other than local autograft bone.
3. There is inadequate tissue coverage over the operative site.
4. There is an open wound local to the operative area, or rapid joint disease, bone absorption, or osteoporosis.
5. Subject has a condition requiring medications that may interfere with bone or soft tissue healing(i.e., oral or parenteral glucocorticoids, immunosuppressives, methotrexate, etc.).
6. Subject has an active local or systemic infection.
7. Subject has a metal sensitivity/foreign body sensitivity (cages will be implanted).
8. Subject is morbidly obese, defined as a body mass index (BMI) greater than 40.
9. Subject has any medical condition or extenuating circumstance that, in the opinion of the investigator, would preclude participation in the study.
10. Subject is currently involved in another investigational drug or device study that could confound study data.
11. There is a history (present or past) of substance abuse (recreational drugs, prescription drugs or alcohol) that in the investigator's opinion may interfere with protocol assessments and/or with the subject's ability to complete the protocol required follow-up.
12. Subjects who are pregnant or plan to become pregnant in the next 12 months or who are lactating. This restriction is due to the inherent risk radiography presents to an embryo or fetus and is considered standard of care.
13. Subject is involved in or planning to engage in litigation or receiving Worker's Compensation related to neck or back pain. Participation may effect the assessments made by case workers and legal teams.
14. Subject is a prisoner.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Brantigan-Steffee-Frasier (BSF) Fusion Scale | Six months following procedure
  Graded radiographic evaluation of ossification and/or pseudarthrosis between vertebrae. The evaluation applies a three-level scale of fusion success:
  BSF-1: Radiographical pseudarthrosis BSF-2: Radiographical locked pseudarthrosis BSF-3: Radiographical fusion
  Radiographic Success: Radiographic success is defined by radiographical fusion (BSF-3) presenting bone bridges within at least half of the fusion area with at least the density originally achieved at surgery.
  Radiographic Failure: Radiographic failure is defined by radiographical pseudarthrosis (BSF-1 or -2)

SECONDARY OUTCOMES:
Oswestry Disability Index (ODIv2.1a) | Preoperative, three, six, twelve, and twenty-four month follow-ups.
  Subject self-assessment survey pertaining to quality-of-life and pain measures. Scale ranges from 0-100%. The higher the percentage, the lower the quality of life and the greater the pain.
Neurological Pain Scale for Back and Legs | Preoperative, three, six, twelve, and twenty-four month follow-ups.
  Subject self-assessment survey pertaining to pain presence in legs and back. The scale runs from 0-10, with 0 indicating no pain and 10 the worst pain possible.
PROMIS-10 Global | Preoperative, three, six, twelve, and twenty-four month follow-ups.
  Patient reported survey to rate quality-of-life and pain experience throughout life of study. Initially gives a raw score for both physical and mental well-being between 4 and 20, which is converted into a T-score between 16.2 and 67.7. The T-score is directly correlated with what is being evaluated. In other words, the higher the T-score, the higher the quality of life and the lower the pain.

CONTACTS AND LOCATIONS:
Overall Officials: Francis Farhadi, MD, PhD, Principal Investigator — University of Kentucky; Craig van Horne, MD, PhD, Study Director — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No